CLINICAL TRIAL: NCT01687569
Title: Effects of Added Spice Flour on Glycaemic Responses to a Cracker Snack
Brief Title: Glycaemic Responses to Cracker Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Reading Scientific Services Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P12-05774
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Glycaemic Response Measurements
Keywords: Glycaemic Response

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Cracker (Placebo Comparator): Base cracker snack
  Interventions: Other: Control Cracker Snack
- Experimental Cracker Snack 1 (Experimental): Cracker snack containing test ingredient 1
  Interventions: Other: Experimental Cracker Snack 1
- Experimental Cracker Snack 2 (Experimental): Cracker snack containing test ingredient 2
  Interventions: Other: Experimental Cracker Snack 2

INTERVENTIONS:
Other: Control Cracker Snack — Base cracker snack
  Arms: Control Cracker
Other: Experimental Cracker Snack 1 — Cracker snack containing test ingredient 1
  Arms: Experimental Cracker Snack 1
Other: Experimental Cracker Snack 2 — Cracker snack containing test ingredient 2
  Arms: Experimental Cracker Snack 2

SUMMARY:
The purpose of this study is to determine whether added ingredient affects glycaemic responses to a cracker snack.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (not less than 40% Male)
* Aged 18 - 55 years
* Non Smokers
* Have a body mass index between 18.5 to 29.99 kg/m2
* Healthy, non-diabetic, no gastric bypass surgery
* Not allergic to wheat, mustard, dairy, or soy
* Have a fasting plasma glucose (finger-stick) <100 mg/dl (<5.5 mmol/L)
* Willing and able to provide written informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Glycaemic Response(s) to cracker snacks as measured by incremental Area Under the Curve (iAUC) | 120 minutes
  The endpoint will be the blood glucose response curve, calculated from the individual glucose measurements. Evaluated by repeated measures ANOVA on incremental AUC measured in capillary blood.

CONTACTS AND LOCATIONS:
Overall Officials: Rungano Munyuki, Principal Investigator — Reading Scientific Services Limited
Locations (1):
- Reading Scientific Services Limited (RSSL), Reading, United Kingdom